CLINICAL TRIAL: NCT02257853
Title: A Randomized Controlled Trial to Determine the Effectiveness of a Stress Reduction Intervention in Caregivers of Allogeneic Hematopoietic Stem Cell Transplant (HSCT) Recipients
Brief Title: Effectiveness of a Stress Reduction Intervention in Caregivers of Allogeneic Hematopoietic Stem Cell Transplant (HSCT) Recipients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 140201; 14-CC-0201
Record Dates: First submitted 2014-10-03; First posted 2014-10-07 (Estimated); Last update posted 2025-09-02 (Actual); Status verified 2025-07-08

CONDITIONS: Stress, Psychological; Caregivers
Keywords: Caregiver Stress; Cancer Caregivers; Yoga-Based Stress Reduction Intervention; HSCT Caregivers
MeSH Terms: conditions — Stress, Psychological; Caregiver Burden

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): No intervention group
- Intervention (Experimental): Receives stress reduction intervention introduction with daily practice
  Interventions: Other: Stress reduction intervention

INTERVENTIONS:
Other: Stress reduction intervention — Gentle chair yoga and breath work
  Arms: Intervention

SUMMARY:
Background:

- People who have an allogeneic hematopoietic stem cell transplant (HSCT) need help as they recover. Being a caregiver can be stressful to the body and mind. Researchers want to find ways to reduce this stress.

Objective:

- To see how a stress reduction intervention affects the stress levels and health of an HSCT caregiver.

Eligibility:

- Adults age 18 and older who plan to be an active caregiver for a person having their first allogeneic HSCT at the NIH Clinical Center. An active caregiver is someone who will be caring for the person from just before admission for the HSCT until at least 6 weeks after.

Design:

* Participants will be put in either the intervention group or the control group.
* All participants will get the usual caregiver education given to all patients and caregivers having a stem cell transplant at the NIH Clinical Center.
* All participants will have 2 study visits. They will give blood samples. They will have health assessments and brief physical exams. They will fill out study questionnaires and have an exit interview.
* The intervention group will get an MP3 player. It will have an audio file with a stress reduction intervention on it. Participants will do this intervention daily. It takes 20 minutes. They will do gentle stretches and breathing exercises. They will get a diary to track their practice.
* The intervention group also will have follow-up phone calls 2 and 4 weeks after their first clinic visit.
* The person getting the HSCT will not be actively involved in the study.
* The study will last about 2 months.

DETAILED DESCRIPTION:
Millions of Americans provide unpaid care for aging or ill family members and friends. Caregiving for an individual with cancer who is undergoing stem cell transplantation is particularly stressful. The stress of caregiving is associated with many disorders, including sleep disturbances, depression, and anxiety. Although there is good evidence that cancer caregivers experience high levels of stress and stress-related symptoms, few interventions studies have been explored to address this concern in this population.

Stress reduction techniques are important skills for individuals to cope with the stress of cancer caregiving. Mindfulness techniques such as yoga and meditation reduce levels of stress and stress-related symptoms in caregivers. However, many caregivers are reluctant to take time away from the patient to attend to their own health and well-being. Few studies have explored yoga-based stress reduction interventions that can be performed at home or at the patient s bedside.

Based upon our past research examining stress and stress-related symptoms in stem cell transplant caregivers, this study is designed to determine preliminary effectiveness of a yoga-based stress reduction intervention in reducing levels of stress in caregivers during allogeneic hematopoietic stem cell transplant (HSCT). In addition, this study will explorefactors associated with change in caregiver stress and symptoms such as demographics, clinical variables, cardiometabolic and inflammatory markers, and health behaviors.

This study will use a prospective randomized control group design to examine the effects of a six-week yoga-based stress reduction intervention on perceived stress in caregivers of allogeneic HSCT patients. Subjects will be accrued to this protocol if they are a caregiver of an individual undergoing allogeneic HSCT at the Clinical Center, NIH, are greater than or equal to 18 years old, able to read English, stand and sit unassisted, raise arms over head without pain, and able to comprehend the investigational nature of the study. A sample of at least 78 caregivers is needed to adequately evaluate the effectiveness of the intervention.

All caregivers will attend the usual care group education provided at the Clinical Center for transplant caregivers. Caregivers randomized to the intervention group will be scheduled for one session with study personnel to receive a 20 minute audio file of gentle chair yoga poses and guided breath awareness, as well as instructions for performing them, and they will be asked to practice daily. Data, in the form of web-based questionnaires, as well as a physical assessment, demographic interview and blood work will be collected from all study participants at baseline (at or near the time of HSCT) and again at the end of the six-week intervention. There will be no long-term follow-up after the intervention period. Questionnaires include: Caregiver Reaction Assessment, Health-Promoting Lifestyle Profile II, Pittsburgh Sleep Quality Index, Freiburg Mindfulness Scale, PROMIS measures of anxiety, applied cognition, depression, positive affect and well-being, Multidimensional Fatigue Symptom Inventory-Short Form and NIH Toolbox measures of loneliness, self-efficacy, and perceived stress. Subjects will participate in an exit interview at the end of the study and the interventionist will complete a log, based on subject diaries, that tracks subject practice, and discrepancy between planned and actual session date and time. Quantitative analysis techniques will be used in this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age greater than or equal to 18 years old
* Ability to comprehend the investigational nature of the study
* Able to read and speak English
* Agrees to participate in the study
* Able to lift arms over head without pain
* Able to sit and stand from a seated position unassisted
* Intends to serve as an active caregiver* for a patient undergoing their 1st allogeneic HSCT at the NIH Clinical Center

EXCLUSION CRITERIA:

* Age less than or equal to 18 years old
* Pregnant or lactating women
* Inability to comprehend investigational nature of study
* Inability to provide informed consent
* Unable to read and speak English
* Does not agree to participate in study or follow study design
* Serving as a paid caregiver for any individual
* Regular practitioner of yoga, meditation or other mind-body practice (definition: taking classes or practicing at least weekly for at least 2 of the past 6 months).
* Physical function limitations that would interfere with intervention

Caregiver participants will be excluded from the biomarker analysis if they have had:

* Glucocorticosteroid treatment in the last 2 months
* Have a recent (within the last 2 months) acute illness or injury
* Have served as a stem cell transplant donor or have taken filgastrim

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2018-11-08 (Actual); Study Completion 2019-02-07 (Actual)

PRIMARY OUTCOMES:
Perceived stress | Pre & 6 Weeks Post
  To examine whether HSCT caregivers participating in a stress reduction intervention demonstrate improvement in certain individual factors (self-efficacy, burden, and mindfulness), psychosocial factors (stress, anxiety, depression, loneliness, positive affect and well-being), behaviors (health behaviors) and symptoms (sleep, fatigue, depression, and cognitive impairment) compared with HSCT caregivers in the control group.

SECONDARY OUTCOMES:
Cardiometabolic factors | Pre & 6 weeks post
Inflammatory cytokines | Pre & 6 Weeks Post
Self-reported symptoms | Pre & 6 weeks post

CONTACTS AND LOCATIONS:
Overall Officials: Lena J Lee, Ph.D., Principal Investigator — National Institutes of Health Clinical Center (CC)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Derived] Lee LJ, Shamburek R, Son H, Wallen GR, Cox R, Flynn S, Yang L, Bevans M, Wehrlen L, Ross A. Effects of a yoga-based stress reduction intervention on stress, psychological outcomes and cardiometabolic biomarkers in cancer caregivers: A randomized controlled trial. PLoS One. 2022 Nov 10;17(11):e0277009. doi: 10.1371/journal.pone.0277009. eCollection 2022. PMID 36355827
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2014-CC-0201.html